CLINICAL TRIAL: NCT04093479
Title: Impact of Maternal BMI on Plasma Levels of Oxytocin During Labor Augmentation
Status: Completed | Type: Observational
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Marie Blomberg, Professor, Linkoeping University
Other Study IDs: 110930ingo
Record Dates: First submitted 2019-09-14; First posted 2019-09-18 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Maternal Obesity During Childbirth; Labor; Arrested Active Phase
Keywords: labor; obesity; oxytocin
MeSH Terms: conditions — Obesity | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — bloodplasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BMI, oxytocin: Repeteadly blood samples will be taken
  Interventions: Other: blood samples

INTERVENTIONS:
Other: blood samples — blood samples will be taken repeatedly

SUMMARY:
The aim of this study is to examine the associations between maternal BMI and levels of oxytocin in maternal plasma during augmentation with oxytocin during first stage of labor in term pregnancy.

DETAILED DESCRIPTION:
A translational prospective experimental study in the delivery ward in Linköping. The study population will include women in two BMI groups (underweight/normal weight and overweight/obese) during first stage of labor with singleton full term pregnancy and cephalic presentation.The BMI is calculated from weight and height registered at the first antenatal visit around week 8-12. At the delivery ward, if the women are in need of labor augmentation with oxytocin infusion, a peripheral venous catheter will be placed in the contralateral arm from the arm where oxytocin will be administrated. The oxytocin infusion will be prepared to a concentration of 10 mU/ml and will be given according to a standardized protocol or to an infusion level giving maximum of 5 uterine contractions per 10 minutes. Blood samples for measuring plasma levels of oxytocin will be taken prior to start and before every increase in the rate of oxytocin infusion. The blood samples will be collected through the first stage of labor.

ELIGIBILITY:
Inclusion Criteria:

Full-term pregnancy (from gestational week 37+0), singel pregnancy, vertex presentation, knowledge in the Swedish language, 18 years and older, known BMI, need of labor augmentation with oxytocin infusion during opening stage.

Exclusion Criteria:

Not participating in other studies at the delivery ward

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Full-term pregnancy (from gestational week 37+0), singel pregnancy, vertex presentation, knowledge in the Swedish language, 18 years and older, known BMI, need of labor augmentation with oxytocin infusion during opening stage.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
maternal BMI, were weight and height will be combined to report BMI in kg/m^2 | eight hours
  mass spectrometry
level of oxytocin in plasma during oxytocin infusion | eight hours
  mass spectrometry

CONTACTS AND LOCATIONS:
Overall Officials: Marie Blomberg, PhD, Principal Investigator — Linkoeping University
Locations (1):
- Department of Obstetrics, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers

REFERENCES:
- [Derived] Ramo Isgren A, Carlhall S, Dennis Retrato M, Kodikara C, A Ubhayasekera K, Kjolhede P, Bergquist J, Blomberg M. The association between maternal body mass index and serial plasma oxytocin levels during labor. PLoS One. 2023 Aug 11;18(8):e0290038. doi: 10.1371/journal.pone.0290038. eCollection 2023. PMID 37566578